CLINICAL TRIAL: NCT03463525
Title: An Open-label PET Study to Determine Brain Exposure of Osimertinib After IV Microdose Administration of [11C]Osimertinib and Therapeutic Oral Doses of Osimertinib to Patients With EGFR Mutated NSCLC With Brain Metastases
Brief Title: Open-label PET Study With [11C]Osimertinib in Patients With EGFRm NSCLC and Brain Metastases
Acronym: ODIN-BM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D5160C00043
Record Dates: First submitted 2018-02-20; First posted 2018-03-13 (Actual); Results first posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2022-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [11C]osimertinib + oral osimertinib (Experimental): IV microdose administrations of [11C]osimertinib co-administered with 80 mg daily oral osimertinib.
  Interventions: Drug: Osimertinib; Drug: [11C]osimertinib

INTERVENTIONS:
Drug: Osimertinib — Osimertinib 80 mg once daily p.o. will be taken continuously by the patient from the day of the second PET exam.
  Other Names: Tagrisso; AZD9291
Drug: [11C]osimertinib — Patients will receive 3 single IV microdose administrations of [11C]osimertinib and PET exams on: Day 1, Day 2 (or up to Day 8) and Day 29.
  Other Names: [11C]AZD9291

SUMMARY:
This is an open-label, single centre, Phase I study to determine the brain exposure of [11C]osimertinib in patients with EGFRm NSCLC with brain metastases.

DETAILED DESCRIPTION:
A Single-centre, Open-label, PET imaging and Pharmacokinetic Study of IV Administered [11C]osimertinib in EGFRm Non-small cell lung cancer patients with brain metastases. The study will consist of 2 phases, an imaging phase and a continuous access phase.

ELIGIBILITY:
Inclusion Criteria

1. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses. Procedures performed for routine clinical practice up to 2 weeks before the provision of written consent are acceptable if not intentionally done for study purposes.

   If a patient declines to participate in any voluntary exploratory research and/or genetic component of the study, there will be no penalty or loss of benefit to the patient and he/she will not be excluded from other aspects of the study.
2. Male or female aged at least 18 years.
3. Histological or cytological confirmation of diagnosis of NSCLC.
4. Confirmation that the tumour harbours an EGFR mutation known to be associated with EGFR-TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q) or T790M EGFR resistance mutation as assessed by local laboratory/or central laboratory via tissue/cytology or in plasma.
5. Mandatory provision (if available) of formalin fixed, paraffin embedded tissue and blood for central confirmation of EGFR mutation status. Please refer to the Laboratory Manual for details.
6. In all patients enrolled, confirmed BM as having at least one non-measurable and/or measurable brain lesion at baseline as per CNS RECIST 1.1 via MRI imaging.
7. World Health Organisation (WHO) performance status 0 to 2 and a minimum life expectancy of 4 weeks.
8. Females should be using adequate contraceptive measures (up to 6 months after the last administration), should not be breastfeeding and must have a negative serum pregnancy test prior to start of dosing if of childbearing potential or must have evidence of non-childbearing potential by fulfilling 1 of the following criteria at screening:

   * Post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments.
   * Women under 50 years old would be consider postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with luteinising hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the institution.
   * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
9. Male subjects should be willing to use barrier contraception
10. Have a body mass index (BMI) between 18.0 kg/m2 and 30.0 kg/m2 inclusive and weigh at least 40.0 kg and no more than 100.0 kg, inclusive
11. Able and willing to participate in all scheduled evaluations, abide by all study restrictions, and complete all required tests and procedures.

Exclusion Criteria

1. Participation in another clinical study with an IP during the previous 14 days (or longer, depending on characteristics of agents used).
2. Treatment with any of the following: EGFR-TKI (e.g. erlotinib, gefitinib or afatinib) within 10 days or at least 5x the half-life, whichever is the longer; any cytotoxic chemotherapy, investigational agents or other anticancer drugs within 14 days of start of IP; osimertinib in the present or other studies; major surgery (excluding placement of vascular access) within 4 weeks of start of IP; radiotherapy (including brain) with a limited field of radiation within 1 week of start of IP, except in patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation which must be completed within 4 weeks of the first administration of the IP; current receipt (or inability to stop at least 3 weeks before study start) medications or herbal supplements known to be potent inducers of CYP3A4.
3. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting the IP with the exception of alopecia and grade 2, prior platinum therapy-related neuropathy.
4. History of brain surgery or major brain trauma in the last year (if the surgery is in the same hemisphere as the brain metastasis).
5. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses or active infection including hepatitis B, hepatitis C and HIV.
6. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) >470 msec obtained from 3 ECGs, using the screening clinic ECG machine derived QTc value.
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (eg, complete left bundle branch block, third degree heart block, second degree heart block).
   * Patient with any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as electrolyte abnormalities including:

     * Serum/plasma potassium <lower limit of normal (LLN)
     * Serum/plasma magnesium <lower limit normal (LLN)
     * Serum/plasma calcium <lower limit normal (LLN)
   * Heart failure, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes.
7. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
8. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   * ANC <1.5 × 109/L; Platelets <100 × 109/L; Haemoglobin <90 g/L;
   * Alanine aminotransferase (ALT) >2.5x ULN or >5x ULN in the presence of liver metastases;
   * Aspartate aminotransferase (AST) >2.5x ULN or >5x ULN in the presence of liver metastases;
   * Total bilirubin >1.5x ULN or >3x ULN in the presence of liver metastases or Gilbert's Syndrome;
   * Creatinine >1.5xl ULN concurrent with creatinine clearance <50 mL/min (using Cockcroft-Gault formula).
9. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the tablet or previous significant bowel resection that would preclude adequate absorption of osimertinib.
10. History of hypersensitivity to active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib.
11. In addition, the following is considered a criterion for exclusion from the exploratory genetic research:

    * Previous allogenic bone marrow transplant
    * Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection
12. Patients on anticoagulant treatment.
13. Absence of collateral flow between ulnar and radial artery as assessed by the Allen´s test".
14. Suffering from claustrophobia and/or having implanted metal devices or implants such as pacemaker, vascular or heart valves or metal deposits such as bullets, shells, metal grains in the eyes.
15. Previous participation in a research PET or PET/CT study.
16. The following are exclusion criteria for contrast enhanced MRIs:

    * Glomerular filtration rate <30 ml/min
    * History of renal insufficiency
    * Pregnancy
17. Women who are breast-feeding.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Ekman, MD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Research Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00043&attachmentIdentifier=3455e587-d5fe-4d36-a5cb-e3f214230eef&fileName=D5160C00043_CSP_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00043&attachmentIdentifier=301d318d-8777-4921-b1bc-bc60764c9b8f&fileName=D5160C00043_CSR_Synopsis_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00043&attachmentIdentifier=127e90f9-272c-425b-a820-bef579c9c191&fileName=D5160C00043_SAP_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 1 study was conducted in participants with epidermal growth factor receptor mutation positive non-small cell lung cancer with brain metastases at a single center in Sweden.
Pre-assignment Details: The study consisted of 2 phases, an Imaging Phase and a Continued Access Phase. A total of 4 participants were enrolled in this study. All 4 participants received treatment and completed the study.
Groups:
- All Participants: Participants received [11C]osimertinib intravenous (IV) microdose (< 10 microgram [μg]) with radioactivity of 300 megabecquerel (MBq)/70 kilogram (kg) of body weight prior to positron emission tomography (PET) examinations on Day 1, Day 2 (or up to Day 8), and Day 25 (±4 days). The minimum injected radioactivity was 200 MBq/70 kg and the maximum was 330 MBq/70 kg of body weight. Additionally, participants received osimertinib 80 milligram (mg) oral tablets once daily from the day of the second PET examination for at least 21 days till the third PET examination.
Period: Overall Study
Arm/Group | All Participants
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least one administration of [11C]osimertinib and/or osimertinib.
Groups:
- All Participants: Participants received [11C]osimertinib IV microdose (< 10 μg) with radioactivity of 300 MBq/70 kg of body weight prior to PET examinations on Day 1, Day 2 (or up to Day 8), and Day 25 (±4 days). The minimum injected radioactivity was 200 MBq/70 kg and the maximum was 330 MBq/70 kg of body weight. Additionally, participants received osimertinib 80 mg oral tablets once daily from the day of the second PET examination for at least 21 days till the third PET examination.
Arm/Group | All Participants
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration of Percent of Injected Dose in the Whole Brain (Cmax, %ID Brain) of [11C]Osimertinib
Description: During the PET examination time, a series of arterial blood samples were taken to measure Cmax, %ID brain of [11C]osimertinib.
Time Frame: Day 1, Day 2 (or up to Day 8) and Day 25
Population: The PET analysis set included all participants who completed at least one PET examination for the evaluation of [11C]osimertinib brain distribution.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent of radioactive drug
Arm/Group | All Participants
Number analyzed (Participants) | 4
percent of radioactive drug
  Day 1: PET1 | 1.465 (9.6)
  Day 2 (or up to Day 8): PET2 | 1.617 (6.6)
  Day 25: PET3 | 1.492 (15.1)

2. Primary Outcome: Maximum Concentration of Brain Standardized Uptake Value (Cmax, SUV Brain) of [11C]Osimertinib
Description: During the PET examination time, a series of arterial blood samples were taken to measure Cmax, SUV brain of [11C]osimertinib.
Time Frame: Day 1, Day 2 (or up to Day 8) and Day 25
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: SUV
Arm/Group | All Participants
Number analyzed (Participants) | 4
SUV
  Day 1: PET1 | 1.006 (27.1)
  Day 2 (or up to Day 8): PET2 | 1.111 (22.0)
  Day 25: PET3 | 1.054 (29.1)

3. Primary Outcome: Time of Maximum Radioactivity Concentration in the Brain (Tmax, Brain) of [11C]Osimertinib
Description: The Tmax, brain was determined directly from the observed concentration versus time data.
Time Frame: Day 1, Day 2 (or up to Day 8) and Day 25
Population: as for outcome 1
Measure: Median (Full Range); unit: minutes
Arm/Group | All Participants
Number analyzed (Participants) | 4
minutes
  Day 1: PET1 | 22.160 [10.67 to 42.23]
  Day 2 (or up to Day 8): PET2 | 36.340 [8.83 to 78.25]
  Day 25: PET3 | 37.125 [16.83 to 60.30]

4. Primary Outcome: Brain to Plasma Partition Coefficient (Kp) of [11C]Osimertinib
Description: The Kp was defined as ratio of radiolabeled drug in brain to that in plasma calculated as area under the brain radioactivity concentration-time curve between 0 and 90 minutes/area under the plasma radioactivity concentration-time curve between 0 and 90 minutes.
Time Frame: Day 1, Day 2 (or up to Day 8) and Day 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | All Participants
Number analyzed (Participants) | 4
ratio
  Day 1: PET1 | 3.753 (0.8328)
  Day 2 (or up to Day 8): PET2 | 3.960 (0.9413)
  Day 25: PET3 | 4.658 (1.5362)

5. Secondary Outcome: Maximum Concentration at Steady State (Css,Max) of Osimertinib and Metabolite AZ5104
Description: Venous blood samples were collected to determine Css,max of osimertinib and metabolite AZ5104.
Time Frame: Pre-dose and 2, 4 and 7.5 hours postdose on Day 25
Population: The Pharmacokinetic (PK) analysis set included all participants who received at least one administration of either [11C]osimertinib and/or osimertinib and had postadministration PK assessments of osimertinib and/or its metabolite AZ5104 without any protocol deviations or administration deviations that could have affected the PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole per liter (nmol/L)
Arm/Group | All Participants
Number analyzed (Participants) | 4
nanomole per liter (nmol/L)
  Osimertinib | 648.0 (29.61)
  Metabolite AZ5104 | 76.53 (59.58)

6. Secondary Outcome: Time of Maximum Drug Concentration at Steady State (Tss,Max) of Osimertinib and Metabolite AZ5104
Description: Venous blood samples were collected to determine tss,max of osimertinib and metabolite AZ5104.
Time Frame: Pre-dose and 2, 4 and 7.5 hours postdose on Day 25
Population: The PK analysis set included all participants who received at least one administration of either [11C]osimertinib and/or osimertinib and had postadministration PK assessments of osimertinib and/or its metabolite AZ5104 without any protocol deviations or administration deviations that could have affected the PK analysis.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | All Participants
Number analyzed (Participants) | 4
hours (h)
  Osimertinib | 4.0 [4.0 to 6.0]
  Metabolite AZ5104 | 4.0 [0.0 to 6.0]

7. Secondary Outcome: Area Under the Concentration-Time Curve at Steady State (AUCss) of Osimertinib and Metabolite AZ5104
Description: Venous blood samples were collected to determine AUCss of osimertinib and metabolite AZ5104.
Time Frame: Pre-dose and 2, 4 and 7.5 hours postdose on Day 25
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | All Participants
Number analyzed (Participants) | 4
h*nmol/L
  Osimertinib | 13080 (32.70)
  Metabolite AZ5104 | 1666 (64.12)

8. Secondary Outcome: Metabolite to Parent Ratio of AUCss
Description: Venous blood samples were collected to determine AUCss of osimertinib and metabolite AZ5104.
Time Frame: Pre-dose and 2, 4 and 7.5 hours postdose on Day 25
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | All Participants
Number analyzed (Participants) | 4
ratio | 0.1274 (27.89)

9. Secondary Outcome: Metabolite to Parent Ratio of Css,Max
Description: Venous blood samples were collected to determine Css,max of osimertinib and metabolite AZ5104.
Time Frame: Pre-dose and 2, 4 and 7.5 hours postdose on Day 25
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | All Participants
Number analyzed (Participants) | 4
ratio | 0.1181 (28.91)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first dose administration of study drug (Day 1) up to 30 days after last dose administration of study drug, approximately 55 days.
Description: The safety analysis set included all participants who received at least one administration of [11C]osimertinib and/or osimertinib.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=4)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Taste disorder (Nervous system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin oedema (Skin and subcutaneous tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic resulted in recruitment being put on hold due to the PET center closing. The Global Study Team endorsed the decision to have fewer participants than anticipated. Participants enrolled in the study continued as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT03463525/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT03463525/SAP_001.pdf